CLINICAL TRIAL: NCT05827094
Title: Pilot Evaluation of a Mobile Intervention to Support Mediterranean Diet (MedD) for Persons With Mild Alzheimer Disease and Alzheimer Disease Related Dementia's (AD/ADRD) and Frailty
Brief Title: Pilot Mobile for Dementia and Frailty
Acronym: Mindful Meals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Oleg Zaslavsky, Associate Professor- School of Nursing, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: STUDY00015813; 5P30DK017047-45 (NIH)
Record Dates: First submitted 2023-04-12; First posted 2023-04-24 (Actual); Results first posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-02

CONDITIONS: Dementia; Frailty
Keywords: Diet; Nutrition; Mediterranean Diet
MeSH Terms: conditions — Dementia; Frailty

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile Intervnetion (Experimental): Participants randomized to the intervention arm will receive verbal and written instructions as well as one-on-one demonstration of the app features. Participants will have an option of either receiving the study mobile device or will be able to use their own device with an installed app. Following the training, participants will be asked to use the app at least once a week.
  Interventions: Other: Mobile app
- Usual Care (Active Comparator): Participants randomly allocated to the control group will receive educational materials on healthy eating, as provided on the NIA web page (https://www.nia.nih.gov/health/healthy-eating).
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Mobile app — The main mobile intervention features. Tracking and immediate feedback: Pressing the icon launches a short series of questions with multiple-choice response options focusing on recent meals . The survey items are modeled after the 14-item Mediterranean Adherence Screener using simplified language and intuitive visuals to lower cognitive load. Based on responses to the survey, the app provides an intuitive visualization of the survey results, personalized feedback, and recipes on how to improve the person's diet. On-demand resources: individuals are able to access on-demand resources about the MedD diet, its benefits, and best dietary practices. The recipe page includes a personalized list of simple breakfast, lunch, dinner, and snack recipes based on the survey results with step by step instructions on how to prepare Mediterranean foods. In-app messaging: Individuals are able to receive notifications and send and receive messages.
  Arms: Mobile Intervnetion
Other: Usual Care — Participants randomly allocated to the control group will receive educational materials on healthy eating, as provided on the NIA web page (https://www.nia.nih.gov/health/healthy-eating).
  Arms: Usual Care

SUMMARY:
In this project, we propose to build on our Stage I formative work (according to the NIH Stage Model for Behavioral Intervention Development), where we developed fully functional prototypes of a mobile intervention aimed at improving adherence to Mediterranean Diet (MedD) for older adults with frailty and early dementia to complete the Stage II exploratory work, where the intervention will undergo further feasibility, acceptability, and preliminary efficacy tests. The intervention includes a patient-facing app that allows users to track their diet and receive personalized feedback concerning opportunities for improvement and recipes for breakfast, lunch, dinner, and snacks, informational materials about MedD, and a chat feature. On the other end, a web-based provider interface allows clinicians to review patient progress, suggest meal plans, and send and receive messages. The pilot randomized controlled trial, conducted over three months, will compare usual care to usual care plus mobile intervention to gather preliminary efficacy data concerning a change in adherence to MedD score (primary outcome). Mechanistic and secondary outcomes will include MedD knowledge, constructs from Social Cognitive Theory (self-efficacy, outcome expectation, self-regulation, and social support), platform use, anthropometric, and functional measures. Feasibility will be evaluated in terms of recruitment and retention outcomes. Acceptability will be determined through post-intervention semi-structured interviews and structured survey measures.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years or older;
2. ICD-9-CM (ICD-10-CM) codes for mild or major neurocognitive disorders with mild-to-moderate severity due to several possible etiologies. Specifically, a) mild neurocognitive disorder 331.83 (G31.84); major neurocognitive disorder 294.1x (F02.8x) due to Alzheimer disease 331.0 (G30.9); frontotemporal lobar degeneration 331.19 (G31.09); Lewy body disease 331.82 (G31.83);
3. mild-to-moderate frailty
4. own a mobile device.

Exclusion Criteria:

1. Severe sensory impairment that makes it impossible to operate a mobile device or respond to prompts
2. English reading level below 6th grade
3. no care partner
4. optimal diet

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Zaslavsky, PhD, MHA, RN, Principal Investigator — University of Washington
Locations (1):
- Univeristy of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Mobile: Were asked to use Mindful Meals mobile app at least once a week
- Control: Received educational materials on healthy eating
Period: Overall Study
Arm/Group | Mobile | Control
Started | 10 | 9
Completed | 9 | 9
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mobile Intervention: Participants randomized to the intervention arm will receive verbal and written instructions as well as one-on-one demonstration of the app features. Participants will have an option of either receiving the study mobile device or will be able to use their own device with an installed app. Following the training, participants will be asked to use the app at least once a week.
  Mobile app: The main mobile intervention features. Tracking and immediate feedback: Pressing the icon launches a short series of questions with multiple-choice response options focusing on recent meals . The survey items are modeled after the 14-item Mediterranean Adherence Screener using simplified language and intuitive visuals to lower cognitive load. Based on responses to the survey, the app provides an intuitive visualization of the survey results, personalized feedback, and recipes on how to improve the person's diet. On-demand resources: individuals are able to access on-demand resources about the MedD diet, its benefits, and best dietary practices. The recipe page includes a personalized list of simple breakfast, lunch, dinner, and snack recipes based on the survey results with step by step instructions on how to prepare Mediterranean foods. In-app messaging: Individuals are able to receive notifications and send and receive messages.
- Total: Total of all reporting groups
Arm/Group | Mobile Intervention | Usual Care | Total
Number analyzed (Participants) | 10 | 9 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 75 (9) | 74 (7) | 74 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 10 | 9 | 19

OUTCOME MEASURES:

1. Primary Outcome: Change in Adherence to Mediterranean Diet (aMed) Score. The Change Was Calculated From Two Time Points as the Value at the Later Time Point Minus the Value at the Earlier Time Point
Description: Mediterranean Diet adherence was measured using an Food Frequency Questionnaire (FFQ) adherence to Mediterranean Diet (aMED) score. The self-administered FFQ asks participants to report the frequency of consumption and portion size of approximately 125-line items over the last 3 months. A series of foods or beverages define each line item. The aMED score was designed to assess adherence to a Mediterranean dietary pattern. aMED scores range from 0 (nonadherence) to 9 (perfect adherence)
Time Frame: Baseline; 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mobile Intervnetion | Usual Care
Number analyzed (Participants) | 10 | 9
score on a scale | 0 (2) | -0.2 (1)

2. Secondary Outcome: Short Physical Performance Battery
Description: The Short Physical Performance Battery (SPPB) is designed to measure functional status and physical performance. The scale is a composite measure assessing walking speed, standing balance, and sit-to-stand performance. The three tests are summed to give a total score, with a maximum of 12 and a minimum of 0, with a higher score indicating higher function.
Time Frame: Baseline; 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Mediterranean Diet Nutrition Knowledge (MDNK) Questionnaire
Description: Items include questions focused on knowledge about foods and nutrients that are important in the MedD.
Time Frame: Baseline; 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Waist Circumference (WC)
Description: WC at the natural waist or narrowest part of the torso will also be measured to the nearest 0.1 cm
Time Frame: Baseline; 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Body Mass Index
Description: Weight to the nearest 0.1 kg and height to the nearest 0.1 cm will be measured and used to compute BMI.
Time Frame: Baseline; 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Social Cognitive Theory
Description: Social-cognitive theory (SCT) mechanistic variables will be measured using the Food Beliefs Survey and modified to focus on MedD
Time Frame: Baseline; 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Mobile | Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/9
Other Adverse Events (participants affected / at risk) | 0/10 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-23): https://cdn.clinicaltrials.gov/large-docs/94/NCT05827094/Prot_SAP_000.pdf